CLINICAL TRIAL: NCT00584974
Title: A Double-Blind, Placebo-Controlled Study Examining The Safety, Efficacy, and Tolerability of SEP-225289 in Subjects With Major Depressive Disorder (Including Atypical and Melancholic Features)
Brief Title: A Safety, Efficacy and Tolerability Study of SEP-225289
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 360-029
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Depressive Disorder, Major
Keywords: Depression; Mental Disorders; Mood Disorders; Depressive Disorder, Major; Dysthymic Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Mental Disorders; Mood Disorders; Dysthymic Disorder | interventions — SEP 225289; Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.5 mg SEP-225289 (Experimental): 0.5 mg SEP-225289
  Interventions: Drug: SEP-225289
- 2.0 mg of SEP-225289 (Experimental): 2.0 mg of SEP-225289
  Interventions: Drug: SEP-225289
- Venlafaxine (Active Comparator): 150 mg Venlafaxine
  Interventions: Drug: Venlafaxine
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SEP-225289 — 0.5 mg SEP-225289
  Arms: 0.5 mg SEP-225289
Drug: SEP-225289 — 2.0 mg SEP-225289
  Arms: 2.0 mg of SEP-225289
Drug: Venlafaxine — 150 mg Venlafaxine
  Other Names: Effexor
  Arms: Venlafaxine
Drug: placebo — Placebo
  Arms: Placebo

SUMMARY:
To determine the safety, efficacy and tolerability of SEP-225289 in subjects with Major Depressive Disorder

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-dummy, multi-center study of the safety, efficacy and tolerability of SEP-225289 in male and female subjects with MDD. Subjects meeting DSM-IV criteria for Melancholic or Atypical Features specifier are eligible for participation. The study will consist of a screening period, which may last up to 2 weeks, an eight week (56 day) double-blind treatment period, a two week (14 day) wash-out, and a one week (7 day) follow up. Total subject participation will be approximately 91 days (13 weeks). This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* The duration of the current episode must be at least 1 month but not longer than 12 months.
* Subjects must have a primary diagnosis of Major Depressive Disorder.
* Subjects must have had at least one previous, diagnosed episode of MDD in the past 5 years.
* MDD must be the condition that was chiefly responsible for motivating the subject to seek treatment.
* Subject is in general good health.

Exclusion Criteria:

* Subject is participating in, has participated in, or plans to participate in any investigational drug study.
* Subject who has donated blood within the last 30 days or plans to donate blood during and 30 days following participation.
* Known failure to respond (in the past 5 years) to two adequate (dose and duration) antidepressant medications with distance mechanisms of action including tricyclics.
* Subjects who have undergone Electroconvulsive Therapy treatment.
* Treatment with fluoxetine, in the 6 weeks before baseline.
* Subject with psychotic disorders, anorexia nervosa, bulimia or post-traumatic stress disorder.
* Subject with a history or presence of bipolar disorder (i.e., current or past history of manic episode).
* Subjects with Obsessive Compulsive Disorder.
* Subjects with a lifetime diagnosis of Panic Disorder.
* Subject received treatment with antidepressants within 2 weeks.
* Subject with lifetime history of suicidal attempts, alcohol dependence or abuse, drug(s) dependence or abuse (excluding nicotine and caffeine) or has a positive urine drug screen.
* Subject has a history of significant risk of suicide or homicide.
* Bereavement - Defined as death of a loved one within 3 months.
* Subject has a documented history of HIV, hepatitis B or hepatitis C.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 523 (Actual)
Dates: Start 2007-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To assess the safety, efficacy and tolerability of SEP-225289 in subjects with Major Depressive Disorder (MDD) | 56 days

SECONDARY OUTCOMES:
To examine the response to SEP-225289 in MDD subjects meeting DSM_IV criteria for atypical and melancholic features | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, CNS, Study Chair — Sumitomo Pharma America, Inc.
Locations (46):
- United States (46):
  - Little Rock, Arkansas
  - Arcadia, California
  - Beverly Hills, California
  - Costa Mesa, California
  - Garden Grove, California
  - Glendale, California
  - Irvine, California
  - Lafayette, California
  - Oceanside, California
  - San Diego, California
  - Upland, California
  - Denver, Colorado
  - New Britain, Connecticut
  - Bradenton, Florida
  - Fort Myers, Florida
  - Jacksonville, Florida
  - Lauderhill, Florida
  - Maitland, Florida
  - North Miami, Florida
  - Sanford, Florida
  - Atlanta, Georgia
  - Smyrna, Georgia
  - Park Ridge, Illinois
  - Lake Charles, Louisiana
  - Boston, Massachusetts
  - Braintree, Massachusetts
  - Flowood, Mississippi
  - Saint Charles, Missouri
  - Clementon, New Jersey
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - New York, New York
  - The Bronx, New York
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Middleburg Heights, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Irving, Texas
  - Midlothian, Virginia
  - Seattle, Washington